CLINICAL TRIAL: NCT03867084
Title: A Phase 3 Double-blinded, Two-arm Study to Evaluate the Safety and Efficacy of Pembrolizumab (MK-3475) Versus Placebo as Adjuvant Therapy in Participants With Hepatocellular Carcinoma and Complete Radiological Response After Surgical Resection or Local Ablation (KEYNOTE-937)
Brief Title: Safety and Efficacy of Pembrolizumab (MK-3475) Versus Placebo as Adjuvant Therapy in Participants With Hepatocellular Carcinoma (HCC) and Complete Radiological Response After Surgical Resection or Local Ablation (MK-3475-937 / KEYNOTE-937)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3475-937; MK-3475-937 (Other: MSD Protocol Number); KEYNOTE-937 (Other: MSD); 194786 (Registry Identifier: JAPAC-CTI); 2022-501971-24-00 (Registry Identifier: EU CT); U1111-1282-6370 (Registry Identifier: UTN); 2018-004800-20 (EudraCT Number)
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Programmed Cell Death 1 (PD-1, PD1); Programmed Cell Death Ligand 1 (PD-L1, PDL1); Checkpoint Inhibitor; Immunotherapy; Adjuvant
MeSH Terms: conditions — Carcinoma, Hepatocellular; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab (Experimental): Participants receive intravenous (IV) pembrolizumab at 200 mg on Day 1 of each 21-day cycle for up to 17 cycles.
  Interventions: Biological: Pembrolizumab
- Placebo (Placebo Comparator): Participants receive IV placebo on Day 1 of each 21-day cycle for up to 17 cycles.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion of Pembrolizumab 200 mg.
  Other Names: KEYTRUDA®; MK-3475
  Arms: Pembrolizumab
Drug: Placebo — IV infusion of 0.9% normal saline.
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of pembrolizumab (MK-3475) versus placebo as adjuvant therapy in participants with hepatocellular carcinoma (HCC) and complete radiological response after surgical resection or local ablation. The primary hypotheses of this study are that adjuvant pembrolizumab is superior to placebo with respect to: 1) recurrence-free survival (RFS) as assessed by blinded independent central review (BICR); and 2) overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of HCC by radiological criteria and/or pathological confirmation.
* Has an eligibility scan (CT of the chest, triphasic CT scan or MRI of the abdomen, and CT or MRI of the pelvis) confirming complete radiological response ≥4 weeks after complete surgical resection or local ablation. Randomization needs to occur within 12 weeks of the date of surgical resection or local ablation.
* Has no radiologic evidence of disease prior to enrollment.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days prior to Cycle 1, Day 1.
* Has a Child-Pugh class A liver score (5 to 6 points) within 7 days prior to Cycle 1, Day 1.
* Has alpha fetoprotein (AFP) concentration lower than 400 ng/mL within 28 days prior to Cycle 1, Day 1.
* Has controlled hepatitis B (Hep B).
* Has recovered adequately from toxicity and/or complications from the local intervention (surgical resection or local ablation) prior to starting study treatment.
* If female, is not pregnant or breastfeeding, and at least one of the following conditions applies: 1) Is not a woman of childbearing potential (WOCBP); or 2) Is a WOCBP and using a contraceptive method that is highly effective or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (a WOCBP must have a negative pregnancy test within 72 hours before the first dose of study treatment).
* If undergoing surgical resection, has submitted a tumor tissue sample during Screening.
* Has adequate organ function.

Exclusion Criteria:

* Has a known additional malignancy that is progressing or has required active antineoplastic treatment (including hormonal) or surgery within the past 3 years.
* Has had esophageal or gastric variceal bleeding within the last 6 months.
* Has clinically apparent ascites on physical examination.
* Has had clinically diagnosed hepatic encephalopathy in the last 6 months.
* Has received local therapy to liver ablation other than with radiofrequency or microwave ablation.
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has dual active Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) infection at study entry.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has known active tuberculosis (TB; Bacillus tuberculosis).
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
* Has received prior systemic anti-cancer therapy for HCC including investigational agents.
* Is receiving any of the following prohibited concomitant therapies:1) Antineoplastic systemic chemotherapy or biological therapy; 2) Immunotherapy not specified in this protocol; 3) Investigational agents other than pembrolizumab; 4) Radiation therapy; 5) Oncological surgical therapy; or systemic glucocorticoids for any purpose other than to modulate symptoms from an AE that is suspected to have an immunologic etiology.
* Has received a live vaccine within 30 days prior to the first dose of study treatment.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to Cycle 1, Day 1.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to Cycle 1, Day 1.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
* Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 959 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Recurrence-Free Survival (RFS) | Up to ~6 years
  RFS is defined as the time from randomization to first documentation of disease recurrence (local, regional, or distant) as assessed by BICR or by pathology consistent with HCC if required per the site's standard of care, or death due to any cause (both cancer and non-cancer causes of death), whichever occurs first.
Overall Survival (OS) | Up to ~8 years
  OS is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Percentage of Participants who Experience an Adverse Event (AE) | Up to ~8 years
  An AE is defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy can be determined.
Percentage of Participants who Discontinue Study Treatment Due to an AE | Up to ~1 year
  An AE is defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy can be determined.
Change from Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Combined Global Health Status (GHS) / Quality of Life (QoL) Scale Score | Baseline and time of last patient reported outcome (PRO) assessment (up to ~5 years)
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to the questions regarding Global Health Status (GHS; "How would you rate your overall health during the past week?") and Quality of Life ("How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1= Very poor to 7=Excellent). The combined score of GHS (Item 29) and QoL (Item 30) is computed by averaging the raw scores of the 2 items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. The change from baseline in GHS (EORTC QLQ-C30 Item 29) and QoL (EORTC QLQ-C30 Item 30) combined score will be reported.
Change from Baseline in EORTC QLQ-C30 Physical Functioning Scale Score | Baseline and time of last PRO assessment (up to ~5 years)
  The EORTC QLQ-C30 is a cancer specific health-related quality of life questionnaire. Participant responses to 5 questions about their physical functioning (Items 1-5) are scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score of items 1 to 5 was computed by averaging the raw scores of the 5 items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. Higher scores indicate better physical functioning. The change from baseline in EORTC QLQ-C30 Physical Functioning (Items 1-5) combined score will be reported.
Change from Baseline in EORTC QLQ-C30 Role Functioning Scale Score | Baseline and time of last PRO assessment (up to ~5 years)
  The EORTC QLQ-C30 is a cancer specific health-related quality of life questionnaire. The role functioning score is based on participant responses to questions scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score was computed by averaging the raw scores of Items 6 and 7 and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. Higher scores indicate better role functioning. The change from baseline in EORTC QLQ-C30 Role Functioning (Items 6 and 7) combined score will be reported.
Change from Baseline in EORTC QLQ-Hepatocellular Carcinoma Module (EORTC QLQ-HCC18) Abdominal Swelling Scale Score | Baseline and time of last PRO assessment (up to ~5 years)
  The EORTC QLQ-HCC18 is an HCC-specific questionnaire, administered in addition to the EORTC QLQ-C30. The abdominal swelling scale score is based on participant responses to questions scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores will be standardized, so that scores range from 0-100. Higher scores indicate more severe symptoms/problems. Change from baseline in the EORTC QLQ-HCC18 abdominal swelling scale score will be reported.
Change from Baseline in EORTC QLQ-HCC18 Fatigue Scale Score | Baseline and time of last PRO assessment (up to ~5 years)
  The EORTC QLQ-HCC18 is an HCC-specific questionnaire, administered in addition to the EORTC QLQ-C30. The fatigue scale score is based on participant responses to questions scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score was computed by averaging the raw scores of the items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. Higher scores indicate more severe symptoms/problems. Change from baseline in the EORTC QLQ-HCC18 fatigue scale score will be reported.
Change from Baseline in EORTC QLQ-HCC18 Pain Scale Score | Baseline and time of last PRO assessment (up to ~5 years)
  The EORTC QLQ-HCC18 is an HCC-specific questionnaire, administered in addition to the EORTC QLQ-C30. The pain scale score is based on participant responses to questions scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score was computed by averaging the raw scores of the items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. Higher scores indicate more severe symptoms/problems. Change from baseline in the EORTC QLQ-HCC18 pain scale score will be reported.
Change from Baseline in European Quality of Life (EuroQoL)-5 Dimensions, 5-level Questionnaire (EQ-5D-5L) Health Utility Score | Baseline and time of last PRO assessment (up to ~5 years)
  The EQ-5D-5L measured health-related outcomes, assessing 5 health state dimensions (mobility, selfcare, usual activities, pain/discomfort, and anxiety/depression) on a 5-point scale from 1 (no problem) to 5 (extreme problems). The EQ-5D-5L also includes a graded (0 to 100) vertical visual analog scale on which the participant rates their general state of health.
Time to Deterioration (TTD) in the EORTC QLQ-C30 Combined GHS / QoL Scale Score | Baseline and time of last PRO assessment (up to ~5 years)
  EORTC QLQ-C30 is a questionnaire to assess QoL of cancer patients. Participant responses to questions on GHS ("How would you rate your overall health during the past week?") and QoL ("How would you rate your overall QoL during the past week?") were scored on a 7-point scale (1= Very poor to 7=Excellent). The combined score of GHS (Item 29) and QoL (Item 30) was computed by averaging raw scores of the 2 items and applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. TTD was defined as the time from baseline to first onset of ≥10-point negative change (decrease) from baseline in GHS-QoL combined score. A longer TTD indicates a better outcome.
TTD in the EORTC QLQ-C30 Physical Functioning Scale Score | Baseline and time of last PRO assessment (up to ~5 years)
  EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to 5 questions about their physical functioning (Items 1 to 5) are scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score of items 1 to 5 was computed by averaging the raw scores of the 5 items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. TTD was defined as the time from baseline to first onset of ≥10-point negative change (decrease) from baseline in physical functioning (Items 1 to 5). A longer TTD indicates a better outcome.
TTD in the EORTC QLQ-C30 Role Functioning Scale Score | Baseline and time of last PRO assessment (up to ~5 years)
  EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to questions about their role functioning (Items 6 and 7) are scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score of Items 6 and 7 was computed by averaging the raw scores of the items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. TTD was defined as the time from baseline to first onset of ≥10-point negative change (decrease) from baseline in physical functioning (Items 6 and 7). A longer TTD indicates a better outcome.
TTD in the EORTC QLQ-HCC18 Abdominal Swelling Scale Score | Baseline and time of last PRO assessment (up to ~5 years)
  The EORTC QLQ-HCC18 is an HCC-specific questionnaire, administered in addition to the EORTC QLQ-C30. The abdominal swelling scale score is based on participant responses to questions scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores will be standardized, so that scores range from 0-100. Higher scores indicate more severe symptoms/problems. The TTD in EORTC QLQ-HCC18 abdominal swelling scale score will be reported, defined as the time to first onset of a ≥10 point decrease from baseline.
TTD in the EORTC QLQ-HCC18 Fatigue Scale Score | Baseline and time of last PRO assessment (up to ~5 years)
  The EORTC QLQ-HCC18 is an HCC-specific questionnaire, administered in addition to the EORTC QLQ-C30. The fatigue scale score is based on participant responses to questions scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score was computed by averaging the raw scores of the items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. Higher scores indicate more severe symptoms/problems. The TTD in EORTC QLQ-HCC18 fatigue scale score will be reported, defined as the time to first onset of a ≥10 point decrease from baseline.
TTD in the EORTC QLQ-HCC18 Pain Scale Score | Baseline and time of last PRO assessment (up to ~5 years)
  The EORTC QLQ-HCC18 is an HCC-specific questionnaire, administered in addition to the EORTC QLQ-C30. The pain scale score is based on participant responses to questions scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score was computed by averaging the raw scores of the items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. Higher scores indicate more severe symptoms/problems. The TTD in EORTC QLQ-HCC18 pain scale score will be reported, defined as the time to first onset of a ≥10 point decrease from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (249):
- United States (24):
  - Banner MD Anderson Cancer Center ( Site 0026), Gilbert, Arizona
  - The University of Arizona Cancer Center - North Campus ( Site 0039), Tucson, Arizona
  - City of Hope Medical Center ( Site 0027), Duarte, California
  - Smilow Cancer Hospital at Yale New Haven ( Site 0042), New Haven, Connecticut
  - Regional Cancer Center ( Site 0054), Fort Myers, Florida
  - Indiana University Simon Cancer Center ( Site 0075), Indianapolis, Indiana
  - University of Iowa ( Site 0067), Iowa City, Iowa
  - James Graham Brown Cancer Center ( Site 0088), Louisville, Kentucky
  - University of Louisville ( Site 0059), Louisville, Kentucky
  - University Medical Center New Orleans ( Site 0014), New Orleans, Louisiana
  - Massachusetts General Hospital ( Site 0062), Boston, Massachusetts
  - Boston Medical Center ( Site 0025), Boston, Massachusetts
  - Beth Israel Deaconess Medical Ctr. ( Site 0033), Boston, Massachusetts
  - University of Massachusetts Worcester ( Site 0017), Worcester, Massachusetts
  - Henry Ford Hospital-GI/Hepatology Research ( Site 0047), Detroit, Michigan
  - University of New Mexico ( Site 0041), Albuquerque, New Mexico
  - North Shore-Long Island Jewish Health System ( Site 0068), Lake Success, New York
  - Miami Valley Hospital South ( Site 0093), Centerville, Ohio
  - University of Cincinnati Medical Center ( Site 0084), Cincinnati, Ohio
  - ProMedica Flower Hospital ( Site 0090), Sylvania, Ohio
  - Stephenson Cancer Center ( Site 0045), Oklahoma City, Oklahoma
  - Vanderbilt Ingram Cancer Center ( Site 0006), Nashville, Tennessee
  - Baylor Scott & White Medical Center - Temple ( Site 0089), Temple, Texas
  - Virginia Mason Medical Center ( Site 0028), Seattle, Washington
- Argentina (7):
  - Hospital Universitario Austral ( Site 0795), Pilar, Buenos Aires
  - Fundación favaloro para la Docencia e Investigación Médica ( Site 0808), Buenos Aires, Buenos Aires F.D.
  - Hospital Provincial del Centenario ( Site 0794), Rosario, Santa Fe Province
  - Hospital Aleman ( Site 0806), Buenos Aires
  - Hospital Italiano ( Site 0793), Buenos Aires
  - Hospital Britanico de Buenos Aires ( Site 0792), Buenos Aires
  - Clinica de nefrologia urologia y enfermedades cardiovasculares ( Site 0802), Santa Fe
- Australia (8):
  - Royal Prince Alfred Hospital AW ( Site 0225), Camperdown, New South Wales
  - Liverpool Hospital ( Site 0226), Liverpool, New South Wales
  - Princess Alexandra Hospital ( Site 0228), Woollongabba, Queensland
  - Royal Adelaide Hospital ( Site 0234), Adelaide, South Australia
  - Monash Health ( Site 0233), Clayton, Victoria
  - St Vincents Hospital Melbourne ( Site 0227), Fitzroy, Victoria
  - Alfred Health ( Site 0230), Melbourne, Victoria
  - Royal Perth Hospital ( Site 0229), Perth, Western Australia
- Belgium (4):
  - University Hospital Antwerp (UZA) ( Site 0374), Edegem, Antwerpen
  - Erasme Hospital ( Site 0376), Brussels, Bruxelles-Capitale, Region de
  - UZ Gent ( Site 0375), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 0377), Leuven, Vlaams-Brabant
- Brazil (11):
  - CIONC - Centro Integrado de Oncologia de Curitiba ( Site 0813), Curitiba, Paraná
  - Hospital de Cancer de Pernambuco ( Site 0815), Recife, Pernambuco
  - Hospital de Clinicas de Porto Alegre ( Site 0824), Porto Alegre, Rio Grande do Sul
  - Clinica de Oncologia Reichow ( Site 0818), Blumenau, Santa Catarina
  - Centro de Novos Tratamentos Itajai - Clinica de Neoplasias Litoral ( Site 0820), Itajaí, Santa Catarina
  - Hospital Paulistano ( Site 0829), São Paulo, São Paulo
  - Instituto COI de Pesquisa Educacao e Gestao ( Site 0825), Rio de Janeiro
  - Instituto do Cancer do Estado de Sao Paulo - ICESP ( Site 0826), São Paulo
  - Real e Benemerita Associacao Portuguesa de Beneficencia ( Site 0828), São Paulo
  - A.C. Camargo Cancer Center ( Site 0827), São Paulo
  - Casa de Saude Santa Marcelina ( Site 0821), São Paulo
- Complex Cancer Center Plovdiv-First Medical Oncology Department ( Site 0982), Plovdiv, Bulgaria
- Canada (3):
  - Nova Scotia Health Authority QEII-HSC ( Site 0208), Halifax, Nova Scotia
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0211), Montreal, Quebec
  - McGill University Health Centre ( Site 0207), Montreal, Quebec
- China (21):
  - Anhui Provincil Hospital South District ( Site 0181), Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences ( Site 0156), Beijing, Beijing Municipality
  - Peking University People's Hospital ( Site 0191), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 0155), Beijing, Beijing Municipality
  - Fujian Provincial Cancer Hospital ( Site 0165), Fuzhou, Fujian
  - 900 Hospital of the Joint ( Site 0197), Fuzhou, Fujian
  - Guangdong General Hospital ( Site 0166), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital ( Site 0172), Guangzhou, Guangdong
  - Wuhan Union Hospital ( Site 0173), Wuhan, Hubei
  - Hubei Cancer Hospital ( Site 0189), Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University ( Site 0167), Changsha, Hunan
  - Hunan Provincial People Hospital ( Site 0192), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 0168), Changsha, Hunan
  - Fudan University Shanghai Cancer Center ( Site 0161), Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University ( Site 0193), Shanghai, Shanghai Municipality
  - Renji Hospital Shanghai Jiaotong University School of Medicine ( Site 0174), Shanghai, Shanghai Municipality
  - Zhongshan Hospital affiliated to Fudan University ( Site 0153), Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi an Jiaotong University ( Site 0164), Xi’an, Shanxi
  - West China Hospital of Sichuan University ( Site 0162), Chengdu, Sichuan
  - Affiliated Tumor Hospital of Xinjiang Medical University ( Site 0157), Ürümqi, Xinjiang
  - Zhejiang Cancer Hospital ( Site 0171), Hangzhou, Zhejiang
- Denmark (3):
  - Herlev Hospital ( Site 0421), Herlev, Capital Region
  - Aarhus Universitets hospital ( Site 0420), Aarhus N, Central Jutland
  - Odense Universitets Hospital ( Site 0422), Odense C, Region Syddanmark
- France (8):
  - HUS Hopital Hautepierre ( Site 0445), Strasbourg, Bas-Rhin
  - Hopital de la Timone ( Site 0442), Marseille, Bouches-du-Rhone
  - CHU Bordeaux Haut-Leveque ( Site 0437), Pessac, Gironde
  - CHU Rangueil ( Site 0441), Toulouse, Haute-Garonne
  - Hopital Beaujon ( Site 0439), Clichy, Hauts-de-Seine
  - CHU Montpellier. ( Site 0443), Montpellier, Herault
  - Hopital Claude Huriez CHRU LILLE ( Site 0440), Lille, Nord
  - Hopital Paul Brousse ( Site 0447), Villejuif, Val-de-Marne
- Germany (13):
  - SLK-Kliniken Heilbronn GmbH ( Site 0460), Heilbronn, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen ( Site 0466), Tübingen, Baden-Wurttemberg
  - Klinikum rechts der Isar der Technischen Universitaet ( Site 0470), Munich, Bavaria
  - Universitaetsklinikum Wuerzburg ( Site 0468), Würzburg, Bavaria
  - Krankenhaus Nord-West GmbH ( Site 0472), Frankfurt am Main, Hesse
  - Universitaetsklinikum Frankfurt ( Site 0467), Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover ( Site 0458), Hanover, Lower Saxony
  - Universitaetsklinikum Koeln ( Site 0463), Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Duesseldorf ( Site 0461), Düsseldorf, North Rhine-Westphalia
  - Staedtisches Klinikum Dresden ( Site 0471), Dresden, Saxony
  - Universitatsklinikum Carl Gustav Carus ( Site 0459), Dresden, Saxony
  - Charite - Campus Virchow Klinikum ( Site 0457), Berlin
  - Universitaetsklinikum Hamburg-Eppendorf ( Site 0469), Hamburg
- Hong Kong (4):
  - Prince of Wales Hospital ( Site 0268), Hong Kong
  - Pamela Youde Nethersole Eastern Hospital ( Site 0271), Hong Kong
  - Queen Mary Hospital ( Site 0267), Hong Kong
  - Tuen Mun Hospital ( Site 0272), Tuenmen
- Hungary (5):
  - Bacs-Kiskun Megyei Korhaz-Onkoradiologiai Kozpont ( Site 0483), Kecskemét, Bács-Kiskun county
  - SZTE Szent-Gyorgyi Albert Klinikai Kozpont ( Site 0482), Szeged, Csongrád megye
  - Somogy Megyei Kaposi Mór Oktató Kórház-Oncology center ( Site 0484), Kaposvár, Somogy County
  - Semmelweis University ( Site 0480), Budapest
  - Debreceni Egyetem Klinikai Kozpont Onkologiai Tanszek ( Site 0481), Debrecen
- Ireland (2):
  - St Vincent's University Hospital ( Site 0498), Dublin
  - Tallaght University Hospital ( Site 0499), Dublin
- Israel (5):
  - Rambam Medical Center ( Site 0524), Haifa
  - Haddassah Medical Organization - Ein Kerem ( Site 0519), Jerusalem
  - Rabin Medical Center ( Site 0520), Petah Tikva
  - Chaim Sheba Medical Center ( Site 0523), Ramat Gan
  - Sourasky Medical Center ( Site 0522), Tel Aviv
- Italy (10):
  - A O U Policlinico di Modena ( Site 0548), Modena, Abruzzo
  - Azienda Ospedaliera Ordine Mauriziano di Torino ( Site 0542), Turin, Piedmont
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia-Cervello ( Site 0547), Palermo, Sicily
  - Istituto Tumori Giovanni Paolo II ( Site 0543), Bari
  - AOU di Bologna Policliico S. Orsola-Malpighi ( Site 0541), Bologna
  - Azienda Ospedaliero Universitaria Careggi ( Site 0549), Florence
  - Fondazione IRCCS Ca' Granda-Ospedale Maggiore Policlinico ( Site 0550), Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 0540), Milan
  - Ospedale del Mare ( Site 0545), Napoli
  - Azienda Ospedaliero Universitaria Pisana ( Site 0546), Pisa
- Japan (22):
  - Ehime University Hospital ( Site 0123), Tōon, Ehime
  - Kurume University Hospital ( Site 0119), Kurume, Fukuoka
  - Hokkaido P.W.F.A.C Sapporo-Kosei General Hospital ( Site 0102), Sapporo, Hokkaido
  - Kanazawa University Hospital ( Site 0111), Kanazawa, Ishikawa-ken
  - Kagawa University Hospital ( Site 0121), Kita-gun, Kagawa-ken
  - Kagawa Prefectural Central Hospital ( Site 0122), Takamatsu, Kagawa-ken
  - Toranomon Hospital Kajigaya ( Site 0109), Kawasaki, Kanagawa
  - Yokohama City University Medical Center ( Site 0110), Yokohama, Kanagawa
  - Kindai University Hospital ( Site 0116), Sayama, Osaka
  - Saitama Medical University Hospital ( Site 0104), Iruma-gun, Saitama
  - Kyorin University Hospital ( Site 0106), Mitaka, Tokyo
  - Musashino Red Cross Hospital ( Site 0107), Musashino, Tokyo
  - Chiba University Hospital ( Site 0103), Chiba
  - National Hospital Organization Kyushu Medical Center ( Site 0118), Fukuoka
  - Hiroshima University Hospital ( Site 0117), Hiroshima
  - University Hospital, Kyoto Prefectural University of Medicine ( Site 0112), Kyoto
  - Japanese Red Cross Osaka Hospital ( Site 0113), Osaka
  - Osaka Metropolitan University Hospital. ( Site 0114), Osaka
  - Saga-Ken Medical Centre Koseikan ( Site 0120), Saga
  - Toranomon Hospital ( Site 0108), Tokyo
  - The University of Tokyo Hospital ( Site 0105), Tokyo
  - Wakayama Medical University Hospital ( Site 0115), Wakayama
- Malaysia (6):
  - Hospital Universiti Sains Malaysia ( Site 0295), Kubang Kerian, Kelantan
  - Gleneagles Penang ( Site 0290), George Town, Pulau Pinang
  - Penang Adventist Hospital ( Site 0289), George Town, Pulau Pinang
  - Institut Kanser Negara - National Cancer Institute ( Site 0294), Putrajaya Wilayah Persekutuan, Putrajaya
  - Sarawak General Hospital ( Site 0293), Kuching, Sarawak
  - University Malaya Medical Centre ( Site 0288), Kuala Lumpur
- New Zealand (2):
  - Christchurch Hospital ( Site 0247), Christchurch, Canterbury
  - Auckland City Hospital ( Site 0246), Auckland
- Oslo Universitetssykehus HF. Ulleval ( Site 0433), Oslo, Norway
- Poland (7):
  - Izerskie Centrum Pulmonologii i Chemioterapii IZER-MED Spolka z o.o. ( Site 0607), Szklarska Poręba, Lower Silesian Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie ( Site 0620), Lublin, Lublin Voivodeship
  - MTZ Clinical Research Sp. z o. o. ( Site 0608), Warsaw, Masovian Voivodeship
  - Copernicus PL Sp. z o.o. ( Site 0603), Gdansk, Pomeranian Voivodeship
  - ID Clinic ( Site 0619), Mysłowice, Silesian Voivodeship
  - SPZOZ MSWIA z Warminsko-Mazurskim Centrum Onkologii w Olsztynie ( Site 0606), Olsztyn, Warmian-Masurian Voivodeship
  - Szpital Wojewodzki im. Mikolaja Kopernika ( Site 0604), Koszalin, West Pomeranian Voivodeship
- Russia (14):
  - Altay Regional Oncology Dispensary ( Site 0919), Barnaul, Altayskiy Kray
  - Siberian Clinical Center of FMBA ( Site 0918), Krasnoyarsk, Krasnoyarsk Krai
  - Krasnoyarsk Regional Clinical Oncological Dispensary ( Site 0648), Krasnoyarsk, Krasnoyarsk Krai
  - Blokhin National Medical Oncology ( Site 0645), Moscow, Moscow
  - City Clinical Hospital 1 na. NI. Pirogov ( Site 0662), Moscow, Moscow
  - First Moscow State Medical University n.a. I.M.Sechenov ( Site 0661), Moscow, Moscow
  - Hadassah Medical-Clinical Research Department ( Site 0920), Moscow, Moscow
  - National Medical Research Radiological Centre ( Site 0660), Moscow, Moscow
  - Privolzhsky District Medical Center ( Site 0655), Nizhny Novgorod, Nizhny Novgorod Oblast
  - Samara Regional Clinical Oncology Center ( Site 0656), Samara, Samara Oblast
  - Road Hospital JSC Russian railways ( Site 0649), Saint Petersburg, Sankt-Peterburg
  - Russian Scientific Center of Radiology and Surgical Technologies ( Site 0665), Saint Petersburg, Sankt-Peterburg
  - City Clinical Oncology Center ( Site 0646), Saint Petersburg, Sankt-Peterburg
  - Tomsk Scientific Research Institute of Oncology ( Site 0657), Tomsk, Tomsk Oblast
- South Korea (7):
  - National Cancer Center ( Site 0314), Goyang-si, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 0313), Seongnam-si, Kyonggi-do
  - Seoul National University Hospital ( Site 0312), Seoul
  - Severance Hospital Yonsei University Health System ( Site 0309), Seoul
  - Asan Medical Center ( Site 0310), Seoul
  - Samsung Medical Center ( Site 0311), Seoul
  - The Catholic University of Korea. Seoul St. Mary s Hospital ( Site 0315), Seoul
- Spain (11):
  - Hospital Universitari Parc Tauli ( Site 0681), Sabadell, Barcelona
  - Hospital Universitario de Donostia ( Site 0671), Donostia / San Sebastian, Gipuzkoa
  - Complejo Hospitalario Universitario de Santiago ( Site 0668), Santiago de Compostela, La Coruna
  - Hospital Universitario Puerta de Hierro ( Site 0678), Majadahonda, Madrid
  - Hospital Central de Asturias ( Site 0667), Oviedo, Principality of Asturias
  - Hospital Universitari Vall d Hebron ( Site 0674), Barcelona
  - Hospital General Universitario Gregorio Maranon ( Site 0676), Madrid
  - Hospital Ramon y Cajal ( Site 0673), Madrid
  - Hospital Universitario La Paz ( Site 0677), Madrid
  - Hospital Universitario Virgen del Rocio ( Site 0670), Seville
  - Hospital Universitario Miguel Servet-Gastroenterology ( Site 0682), Zaragoza
- Sweden (4):
  - Skane University Hospital ( Site 0692), Malmo, Skåne County
  - Karolinska Universitetssjukhuset, Huddinge ( Site 0689), Stockholm, Stockholm County
  - Norrlands Universitetssjukhus ( Site 0687), Umeå, Västerbotten County
  - Sahlgrenska Universitetssjukhuset ( Site 0691), Gothenburg, Västra Götaland County
- Switzerland (7):
  - Universitaetsspital Bern ( Site 0710), Bern, Canton of Aargau
  - University Hospital Basel ( Site 0709), Basel, Canton of Basel-City
  - Kantonsspital St. Gallen ( Site 0708), Sankt Gallen, Canton of St. Gallen
  - CHUV (centre hospitalier universitaire vaudois) ( Site 0712), Lausanne, Canton of Vaud
  - Kantonsspital Winterthur ( Site 0714), Winterthur, Canton of Zurich
  - Hopitaux Universitaires de Geneve HUG ( Site 0711), Geneva
  - Universitaetsspital Zurich ( Site 0713), Zurich
- Taiwan (6):
  - Chang Gung Medical Foundation. Kaohsiung Branch ( Site 0335), Kaohsiung City
  - China Medical University Hospital ( Site 0333), Taichung
  - National Cheng Kung University Hospital ( Site 0334), Tainan
  - National Taiwan University Hospital ( Site 0330), Taipei
  - Taipei Veterans General Hospital ( Site 0331), Taipei
  - Chang Gung Medical Foundation. Linkou ( Site 0332), Taoyuan District
- Thailand (4):
  - Ramathibodi Hospital. ( Site 0352), Bangkok, Bangkok
  - Siriraj Hospital ( Site 0351), Bangkok, Bangkok
  - Maharaj Nakorn Chiangmai Hospital ( Site 0353), Chiang Mai
  - Srinagarind Hospital ( Site 0354), Khon Kaen
- Turkey (Türkiye) (12):
  - Namik Kemal Universitesi Tip Fakultesi ( Site 0738), Tekirdağ, Tekirdas
  - Baskent Unv. Adana Uyg. ve Arast. Hastanesi ( Site 0733), Adana
  - Gulhane Egitim ve Arastirma Hastanesi ( Site 0741), Ankara
  - Ankara Sehir Hastanesi ( Site 0731), Ankara
  - Adnan Menderes University Medical Faculty ( Site 0737), Aydin
  - Bezmialem Vakif University School of Medicine ( Site 0732), Istanbul
  - Acıbadem Maslak Hastanesi ( Site 0742), Istanbul
  - Göztepe Prof. Dr. Süleyman Yalçın Şehir Hastanesi-oncology ( Site 0730), Istanbul
  - Dokuz Eylul Universitesi ( Site 0740), Izmir
  - Konya Necmettin Erbakan University Medical Faculty ( Site 0736), Konya
  - Inonu University Faculty of Medicine ( Site 0729), Malatya
  - VM Medical Park Hastanesi ( Site 0739), Mersin
- Ukraine (8):
  - Regional Clinical Onco Dispensary_ State Medical University ( Site 0782), Chernivtsi, Chernivetska Oblast
  - Regional Oncology Center of Kharkiv ( Site 0777), Kharkiv, Kharkivs’ka Oblast’
  - National Cancer Institute of the MoH of Ukraine ( Site 0779), Kyiv, Kyivska Oblast
  - Shalimov s NI of Surgery and Transplantation ( Site 0781), Kyiv, Kyivska Oblast
  - MI Odessa Regional Oncological Centre ( Site 0776), Odesa, Odesa Oblast
  - CI City Clinical Hospital # 3 ( Site 0783), Zaporizhzhia, Zaporizhzhia Oblast
  - Universal Clinic Oberig-Oncology Center ( Site 0786), Kyiv
  - Medical Center Dobrobut Clinic ( Site 0785), Kyiv
- United Kingdom (9):
  - Cambridge University Hospitals NHS Trust ( Site 0755), Cambridge, Cambridgeshire
  - Weston Park Hospital ( Site 0753), Sheffield, Derbyshire
  - The Beatson West of Scotland Cancer Centre ( Site 0750), Glasgow, Glasgow City
  - Kings College Hospital NHS Foundation Trust ( Site 0758), London, London, City of
  - Belfast City Hospital ( Site 0752), Belfast, Northern Ireland
  - The Clatterbridge Cancer Centre NHS Foundation Trust ( Site 0757), Birkenhead, Wirral
  - University Hospital Coventry and Warwickshire NHS Trust ( Site 0754), Coventry
  - Leeds Teaching Hospitals NHS Trust ( Site 0751), Leeds
  - Nottingham University Hospitals NHS Trust ( Site 0756), Nottingham

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Verset G, Borbath I, Karwal M, Verslype C, Van Vlierberghe H, Kardosh A, Zagonel V, Stal P, Sarker D, Palmer DH, Vogel A, Edeline J, Cattan S, Kudo M, Cheng AL, Ogasawara S, Daniele B, Chan SL, Knox JJ, Qin S, Siegel AB, Chisamore M, Hatogai K, Wang A, Finn RS, Zhu AX. Pembrolizumab Monotherapy for Previously Untreated Advanced Hepatocellular Carcinoma: Data from the Open-Label, Phase II KEYNOTE-224 Trial. Clin Cancer Res. 2022 Jun 13;28(12):2547-2554. doi: 10.1158/1078-0432.CCR-21-3807. PMID 35421228
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26207&tenant=MT_MSD_9011